CLINICAL TRIAL: NCT06616766
Title: A Phase 1/2, Open-label, Multicenter, FIH Study to Evaluate the Safety, Tolerability, PK and Anti-tumor Activity of YH42946 in Patients With Locally Advanced or Metastatic Solid Tumors With HER2 Aberration and EGFR Exon 20 Insertion
Brief Title: A Phase 1/2, Open-label, Multicenter, FIH Study to Evaluate Safety, Tolerability, PK and Anti-tumor Activity of YH42946
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Yuhan Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: YH42946-101
Record Dates: First submitted 2024-09-23; First posted 2024-09-27 (Actual); Last update posted 2025-11-04 (Actual); Status verified 2025-11

CONDITIONS: NSCLC (Non-small Cell Lung Cancer); Solid Tumor
Keywords: YH42946-101
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Part 1 and Part 2 (Experimental): Part 1: Dose escalation arm to determine the MTD Part 2: Dose expansion part to select RD. Several independent cohorts are planned.
  Interventions: Drug: YH42946

INTERVENTIONS:
Drug: YH42946 — YH42946

SUMMARY:
The goal of this YH42946-101 is to evaluate the safety, Tolerability, Pharmacokinetics and anti-tumor activity of YH42946 in patients with locally advanced of metastatic solid tumors with HER2 aberration and EGFR exon 20 insertions.

DETAILED DESCRIPTION:
YH42946 is a novel, orally available tyrosine kinase inhibitor targeting HER2. YH42946 showed potency for diverse HER2 aberrations including HER2 overexpression, amplification, or mutation, as well as EGFR Ex20ins.

This is a Phase 1/2, open-label, multicenter, first-in-human study of YH42946. The study has 2 parts. The first part is dose escalation part to identify the maximum tolerated dose. The second part is dose expansion part to select 2 doses for RD selection at the first cohort, after then RD will be determined to ensure its efficacy. Several independent cohorts are planned.

ELIGIBILITY:
Inclusion Criteria:

* ECOG performance status 0 or 1
* Estimated life expectancy of at least 3 months
* Patients who have progressed on or after all available standard therapies or for whom standard treatment is inappropriate
* Mandatory provision of archived or fresh tumor tissue in quantity sufficient to allow for retrospective confirmation of HER2 or EGFR mutation
* A patient with a history of brain metastases must have had all lesions treated
* Adequate organ function defined as all of the following:

  * Adequate bone marrow function (within 1 week prior to first administration): Neutrophils≥1.5 x10*9 cells/L (Criteria must be met without the use of Granulocyte-Colony Stimulating Factor (G-CSF) within last week prior to testing.); platelet count≥75 x10*9 cells/L; Hb ≥9g/dL (Criteria must be met without packed red blood cell (pRBC) transfusion within last week prior to testing.)
  * Adequate hepatic function: Serum bilirubin≤1.5 x upper limit of normal (ULN), and serum transaminase (either aspartate transaminase (AST) or alanine transaminase (ALT)) ≤ 3 x ULN if no demonstrable liver metastases, or otherwise ≤ 5 x ULN if transaminase elevation is attributable to liver metastases (within 1 week prior to first administration)
  * Adequate renal function: Serum creatinine ≤ 1.5 x ULN or Estimated glomerular filtration rate (eGFR) > 60 mL/min per 1.73 m*2 according to the site's calculation method.

[Dose Escalation part only]

* Histologically or cytologically confirmed diagnosis of advanced, and/or metastatic non-hematologic malignancy
* Documented HER2 or EGFR mutation (HER2 mutation or EGFR exon 20 insertion, HER2 amplification or overexpression)

[Dose Expansion part only]

* Patients with histologically or cytologically confirmed locally advanced or metastatic NSCLC HER2 exon 20 insertion (Cohort 1)

Exclusion Criteria:

* Patient with symptomatic or progressive brain metastases
* Known or suspected leptomeningeal disease (LMD)
* Uncontrolled spinal cord compression
* History of acute coronary syndromes, including myocardial infarction, coronary artery bypass graft, unstable angina, coronary angioplasty or stenting within past 24 weeks
* History of or current Class II, III or IV heart failure as defined by the New York Heart Association (NYHA) functional classification system
* Medical, psychiatric, cognitive or other conditions that compromise the patients ability to understand the patient information, to give informed consent, to comply with the study protocol or to complete the study
* Any severe concurrent disease or condition (includes active infections, cardiac arrhythmia) that in the judgment of the Investigator would make study participation inappropriate for the patient
* History of (non-infectious) interstitial lung disease (ILD) or pneumonitis that required steroids, or any evidence of current ILD or pneumonitis
* History of a second primary cancer with the exception of

  1. curatively treated non-melanomatous skin cancer,
  2. curatively treated cervical or breast carcinoma in situ, or
  3. other malignancy with no known active disease present and no treatment administered during the last 2 years
* Infection with human immunodeficiency virus (HIV) or prior hepatitis B or active chronic hepatitis B or active hepatitis C
* Major surgery within 4 weeks prior to the first dose of study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 161 (Estimated)
Dates: Start 2024-10-02 (Actual); Primary Completion 2028-03-15 (Estimated); Study Completion 2028-07-29 (Estimated)

PRIMARY OUTCOMES:
Treatment Emergent Adverse Events(TEAE)s | Through study completion, during the first 21 days of DLT evaluation period.
  To assess the safety and tolerability of YH42946
Objective Response Rate (ORR) | Through dose expansion part completion, approximately 12 months
  Anti-tumor activity according to RECIST v1.1

SECONDARY OUTCOMES:
AUClast | Through study completion, approximately 12 months
  To characterize the pharmacokinetics (PK) of YH42946
AUCinf | Through study completion, approximately 12 months
  To characterize the pharmacokinetics (PK) of YH42946
Cmax | Through study completion, approximately 12 months
  To characterize the pharmacokinetics (PK) of YH42946
Tmax | Through study completion, approximately 12 months
  To characterize the pharmacokinetics (PK) of YH42946
Objective Response Rate (ORR) | Through study completion, approximately 12 months
  To assess the anti-tumor activity according to RECIST v1.1

OTHER OUTCOMES:
Overall survival(OS) | Through study completion, approximately 3.5 year
  To assess the overall survival of YH42946

CONTACTS AND LOCATIONS:
Overall Officials: Judith Ertle, MD, Study Director — Yuhan Corporation
Locations (8):
- Next Oncology Virginia, Fairfax, Virginia, United States
- South Korea (7):
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - The Catholic Univ. of Korea St. Vincent's Hospital, Suwon, Gyeonggi-do
  - Chungbuk National University Hospital, Cheongju-si, North Chungcheong
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University, Seoul
  - Samsung Medical Center, Seoul
  - Asan Medical Center, University of Ulsan, Seoul

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (including data dictionaries) that underline the results reported in study-related publications will be made available during the period beginning 1 year and ending 5 years after all trial primary and secondary endpoints were assessed. Only requests from researchers who provide a methodologically sound proposal will be reviewed and approved by the sponsor. The analysis type should be in accordance with aims in the proposal approved by the sponsor. Proposals should be directed to clinicaltrials@yuhan.co.kr
  A summary of the study results will be posted in the publicly accessible database (i.e. clinicaltrials.gov) no later than 1 year after the study's primary completion date.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Beginning 1 year and ending 5 years after all trial endpoints were assessed
Access Criteria: Only requests from researchers who provide a methodologically sound proposal will be reviewed and approved by the sponsor. The analysis type should be in accordance with aims in the proposal approved by the sponsor. Proposals should be directed to clinicaltrials@yuhan.co.kr